CLINICAL TRIAL: NCT02464982
Title: Areola Tattoo: the End of a Long Therapeutic Process. A Patient's Quality of Life Dedicated Technology
Brief Title: Psycho-esthetic Impact of Tattoo Technology as Part of Mammary Reconstruction After Surgery Against Breast Cancer
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: PHRIP 2011 / 1 AMC
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Breast Cancer; Right or Left Breast Mammary Reconstruction; Malignant Neoplasm Reconstruction by Tattoo of Areola of Female Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Tattooing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women with 1 year non-invasive technology areola tattoo: Women with 1 year non-invasive technology areola tattoo realized in standard care as part of 1 breast mammary reconstruction following an operated breast cancer
  Interventions: Procedure: Tattoo

INTERVENTIONS:
Procedure: Tattoo — tattoo device with EC standards, and sterile single-use only needle

SUMMARY:
Mammary reconstruction replaces total skin transplant, which may causing patient discomfort. It is a simple, painless and reproductible technology that avoids consequences and complications related to transplant. Tattoo helps patients to return faster to the normal life and close more easily the cancer episode.

The study purpose is to measure the patient's esthetic satisfaction degree on 1year areola tattoo realized following standard care.

DETAILED DESCRIPTION:
Tattoo is realized as standard car as part of mammary reconstruction after surgery of patient suffering from breast cancer. We try to measured :

* Tattooed patient's satisfaction degree with qualitative questionnaire using four level satisfaction scale (very satisfied, satisfied, dissatisfied, very dissatisfied)
* Evaluate from patient and jury, the tall, form, color and areola position defects
* Evaluate professional jury's satisfaction degree regarding this areola tattoo technology, with the same patient criteria

ELIGIBILITY:
Inclusion Criteria:

* technology areola tattoo realized as part of 1 breast mammary reconstruction following an operated breast cancer

Exclusion Criteria:

* Two breasts operated patient
* surgical reconstruction

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women with 1 year non-invasive technology areola tattoo realized as part of 1 breast mammary reconstruction following an operated breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2012-02; Primary Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Patient's satisfaction degree with qualitative questionnaire about them areola tattoo realized after surgery as part of breast cancer treatment | 1 year after areola tattoo have been realized following standard care

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie DUGUET, Principal Investigator — esthetic, reconstruction and maxillo-facial surgery department, University Hospital, Strasbourg
Locations (1):
- esthetic, reconstruction and maxillo-facial surgery department, University Hospital, Strasbourg, France